CLINICAL TRIAL: NCT06864338
Title: Pilot Study for Colorectal Cancer and Advanced Adenoma Detection With the Mainz Biomed Colorectal Cancer Test (eAArly DETECT)
Brief Title: Pilot Study for Colorectal Cancer and Advanced Adenoma Detection With the Mainz Biomed Colorectal Cancer Test
Acronym: eAArly DETECT
Status: Recruiting | Type: Observational
Sponsor: Mainz Biomed (Industry)
Responsible Party: Sponsor
Other Study IDs: MNZ-CRC-002
Record Dates: First submitted 2025-03-03; First posted 2025-03-07 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-06

CONDITIONS: Colorectal Cancer Screening; Colorectal Cancer Metastatic; Colon Adenocarcinoma
Keywords: Stool test; Colorectal cancer screening test; advanced adenoma screeing test
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Individuals aged 45 and over at average risk of colorectal cancer.: Individuals aged 45 and older that are advised to have or are scheduled for a screening colonoscopy and are at average risk for colorectal cancer.
- Individuals aged 18 and older suspected or known to have at least one precancerous, intact lesion.: Individuals aged 18 and older that are suspected to have at least one advanced precancerous lesion or colorectal cancer. Subjects in this group are those that have been pre-identified with imaging, a positive non-invasive screening test, and/or colonoscopy which requires additional intervention.

SUMMARY:
The Mainz Biomed Colorectal Cancer Screening Test is being studied for its performance in the identification of the presence of colorectal cancer (CRC) or advanced adenoma (AA) in the colon in patients at average risk for colorectal cancer.

DETAILED DESCRIPTION:
The primary objectives of this study are:

1. Feasibility and test optimization for the Mainz Biomed Colorectal Cancer Screening Test.
2. To develop the test algorithm and establish the clinical cut-off values for the Mainz Biomed Colorectal Cancer Screening Test.

Each enrolled participant will be asked to provide a stool sample. The stool sample will be shipped to a laboratory and tested. No results will be provided to the site or the participant.

ELIGIBILITY:
Group 1: Screening Group Inclusion Criteria

1. Subject is any sex and ≥45 years of age
2. Subject must be advised to have or be scheduled for a screening colonoscopy
3. Subject is at average risk for colorectal cancer according to the United States Preventive Services Task Force (USPSTF) guidelines, including:

   * no prior diagnosis of colorectal cancer, adenomatous polyps, or inflammatory bowel disease
   * no family history of colorectal cancer (defined as one or more first degree relatives including parent, sibling, or child)
   * no personal diagnosis or family history of known genetic disorders that predispose them to a high lifetime risk of colorectal cancer including:

     * Inflammatory bowel disease (IBD) including chronic ulcerative colitis (CUC) and Crohn's disease
     * Familial adenomatous polyposis (also referred to as "FAP", including attenuated FAP)
     * Hereditary non-polyposis colorectal cancer syndrome (also referred to as "HNPCC" or "Lynch Syndrome")
     * Other hereditary cancer syndromes including but are not limited to Peutz-Jeghers Syndrome, MYH-Associated Polyposis (MAP), Gardner's Syndrome, Turcot's (or Crail's) Syndrome, Cowden's Syndrome, Juvenile Polyposis, Neurofibromatosis and Familial Hyperplastic Polyposis
     * Cronkhite Canada Syndrome
4. Subject can understand the study procedures, and is able to provide consent to participate in the study and authorizes release of relevant protected health information through reviewing and consenting to a Health Insurance Portability and Accountability Act (HIPAA) medical release form
5. Subject is able and willing to provide stool samples within ninety (90) days before the colonoscopy procedure
6. Subject is able and willing to undergo a colonoscopy after providing a stool sample Exclusion Criteria

1. Subject had any precancerous findings on most recent colonoscopy. This does not include non-neoplastic polyps and/or hyperplastic polyps of any size (Note: tissue biopsies that result in no histopathology findings are acceptable) 2. Subject has a history of abnormal imaging suggesting colorectal cancer (e.g., colonography, MRI, CT, barium enema) 3. Subject has a history of any of the following cancers: oral, head and neck, lung, esophagus, gastric, biliary/liver, pancreatic, small bowel, or appendiceal 4. Subject has had a positive non-invasive screening diagnostic within the associated recommended intervals

* High-sensitivity fecal occult blood test or fecal immunochemical test within the previous twelve (12) months
* sDNA-FIT test within the previous thirty-six (36) months 5. Subject has had a colonoscopy in the previous nine (9) years (not including failed/ aborted colonoscopy e.g., due to failed preparation, inability to reach the cecum, patient instability during the procedure, etc.) 6. Subject has had a prior colorectal resection for any reason other than sigmoid diverticular disease 7. Indication for colonoscopy due to overt rectal bleeding (e.g., hematochezia or melena) within the previous thirty (30) days (Note: blood on toilet paper, after wiping, does not constitute rectal bleeding) 8. Subject has any condition that in the opinion of the investigator should preclude participation in the study

Group 2: Diagnostic Group Inclusion Criteria

1. Subject is any sex and ≥ 18 years of age
2. Subject is able and willing to give informed consent
3. Through imaging, a positive non-invasive screening test, or colonoscopy requiring additional intervention subject is suspected or known to have Colorectal Cancer or Advanced Adenoma
4. Subject has not yet been treated (e.g., ablation, surgical resection, radiation, chemotherapy, etc.) and still has at least one intact or partially intact lesion
5. Subject must have a diagnostic colonoscopy or surgical intervention scheduled within 90 days of sample collection
6. Subject can understand the study procedures and is able to provide consent to participate in the study and authorizes release of relevant protected health information through reviewing and consenting to a Health Insurance Portability and Accountability Act (HIPAA) medical release form
7. Subject is able and willing to provide stool samples within ninety (90) days of enrollment and before any treatment procedures are initiated Exclusion Criteria

1. Subject has had a tumor or malignancy other than colorectal cancer identified within the past five years (does not include non-melanoma skin cancer) 2. Subject has been previously diagnosed with inflammatory bowel disease (ulcerative colitis or Crohn's disease) 3. Subject has any condition that in the opinion of the investigator should preclude participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Two groups will be enrolled. Group 1: Screening group at average risk of colorectal cancer. Group 2: Group that has a suspected or known precancerous lesion or colorectal cancer.
Sampling Method: Non-Probability Sample
Enrollment: 2700 (Estimated)
Dates: Start 2022-12-18 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility, test optimization, algorithm, and cut off ranges for the Mainz Biomed Colorectal Cancer Screening Test. | 3 years
  Test results will be used for the feasibility, test optimization, algorithm, and cut- off ranges for the Mainz Biomed Colorectal Cancer Screening Test.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Bresalier, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- Virtual Research Group, Morrisville, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No